CLINICAL TRIAL: NCT04279223
Title: Does Using a 5 mm Telescope in Laparoscopic Cholecystectomy Reduce the Incidence of Trocar Site Hernia? Multicentric Prospective Randomized Study
Brief Title: Does Using a 5 mm Telescope in Laparoscopic Cholecystectomy Reduce the Incidence of Trocar Site Hernia?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Alpaslan Şahin, MD, General Surgeon, Konya Meram State Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Konya TRH General Surgery
Record Dates: First submitted 2020-02-18; First posted 2020-02-21 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Cholelithiasis
MeSH Terms: conditions — Cholelithiasis | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5 mm trocar group (Active Comparator): A study with 107 patients was planned to compare the development of trocar site hernia.
  Interventions: Procedure: Laparoscopic cholecystectomy
- 10 mm trocar group (Sham Comparator): A study with 107 patients was planned to compare the development of trocar site hernia.
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — Comparative study to investigate the effect of small-scale trocar use on the development of trocar site hernia in laparoscopic cholecystectomy

SUMMARY:
10 mm telescope is generally used in laparoscopic cholecystectomy surgery. The use of a 10 mm telescope, although rare, causes the development of a trocar site hernia. İnvestigators thought that the incidence of trocar site hernia would decrease by using a 5 mm trocar, and investigators planned a study.

DETAILED DESCRIPTION:
10 mm telescope is generally used in laparoscopic cholecystectomy surgery. The use of a 10 mm telescope, although rare, causes the development of a trocar site hernia. Investigators thought that the incidence of trocar site hernia would decrease by using a 5 mm trocar, and investigators planned a study.

Elective laparoscopic with a diagnosis of symptomatic cholelithiasis Patients hospitalized in Mogadishu-Somalia Recep Tayyip Erdoğan Training and Research Hospital and Konya Training and Research Hospital General Surgery clinic for cholecystectomy operation will be included in the study and randomized into two groups. In the first group, a 10 mm telescope will be used, and in the second group, a 5 mm telescope will be used. Patients will be followed up for a total of 3 years in 6-month periods for the development of trocar site hernia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic gallstones above 18 years of age

Exclusion Criteria:

* Those with a history of abdominal surgery,
* Open cholecystectomy,
* Patients who develop cholecystectomy complications,
* Those with decompensated systemic disease,
* Patients who do not want to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
Rate of people developing trocar site hernia | Three years has been designed from the completion of the operations.
  Patients in both groups will undergo a physical examination every six months postoperatively. Those with suspected clinical hernia will be evaluated by ultrasonography. Whether the Trokar site hernia has developed will be recorded in the study registration forms. At the end of the third year, the controls will be completed, and the study will be terminated.

CONTACTS AND LOCATIONS:
Overall Officials: alpaslan şahin, md, Study Director — general surgeon
Locations (1):
- Konya Training and Research Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chatzimavroudis G, Papaziogas B, Galanis I, Koutelidakis I, Atmatzidis S, Evangelatos P, Voloudakis N, Ananiadis A, Doundis A, Christoforidis E. Trocar site hernia following laparoscopic cholecystectomy: a 10-year single center experience. Hernia. 2017 Dec;21(6):925-932. doi: 10.1007/s10029-017-1699-3. Epub 2017 Oct 25. PMID 29071498
- [Background] Casaccia M, Papadia FS, Palombo D, Di Domenico S, Sormani MP, Batistotti P, Mascherini M, De Cian F. Single-Port Versus Conventional Laparoscopic Cholecystectomy: Better Cosmesis at the Price of an Increased Incisional Hernia Rate? J Laparoendosc Adv Surg Tech A. 2019 Sep;29(9):1163-1167. doi: 10.1089/lap.2019.0374. Epub 2019 Jul 2. PMID 31264921
- [Background] Hoyuela C, Juvany M, Guillaumes S, Ardid J, Trias M, Bachero I, Martrat A. Long-term incisional hernia rate after single-incision laparoscopic cholecystectomy is significantly higher than that after standard three-port laparoscopy: a cohort study. Hernia. 2019 Dec;23(6):1205-1213. doi: 10.1007/s10029-019-01969-x. Epub 2019 May 9. PMID 31073959